CLINICAL TRIAL: NCT06732908
Title: Evaluating the Safety and Tolerability of LipoMicel Berberine
Brief Title: Safety Profile of a New Berberine Formulation with Improved Bioavailability
Acronym: Berberine Safe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2022-11-002
Record Dates: First submitted 2024-11-28; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Safety
Keywords: berberine; LipoMicel; safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Berberine LipoMicel (Active Comparator): 1000 mg of LipoMicel Berberine (2 soft gel capsules) administered daily to randomized healthy participants for 30 days.
  Interventions: Dietary Supplement: LipoMicel Berberine
- Placebo (Placebo Comparator): Placebo capsules containing microcrystalline cellulose administered daily to randomized healthy participants for 30 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: LipoMicel Berberine — Berberine powder in a LipoMicel matrix encapsulated in soft gel.
  Arms: Berberine LipoMicel
Other: Placebo — microcrystalline cellulose
  Arms: Placebo

SUMMARY:
This study aims to evaluate important safety markers related to liver- and kidney function in healthy individuals after treatment with a new formulation, LipoMicel Berberine. The main question this research aims to answer is:

Is the new formulation of Berberine (LipoMicel) with improved bioavailability safe and well tolerated in healthy individuals?

Participants will:

1. Take 1000 mg (2 capsules/d) of LipoMicel Berberine orally for a maximum period of 30 days.
2. Return to study site weekly for blood tests.
3. Keep a diary of their symptoms (collection of adverse events).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between 21-65 years of age.
* Completed an online health questionnaire on their medical history
* A voluntarily signed informed consent form.

Exclusion Criteria:

* Use of anti-inflammatory or non-steroidal anti-inflammatory medication
* Presence of cardiovascular disease and/or other acute or chronic diseases (e.g., liver, kidney or gastrointestinal diseases).
* Use of cannabis, nicotine or tobacco
* Drinking of excess alcohol (>20 g/day)
* Those who are or plan to become pregnant
* Use of antioxidant supplements
* Use of cholesterol-lowering agents
* Participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Safety of LipoMicel Berberine - ALT | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in liver function based on ALT.
Safety of Lipomicel Berberine - AST | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in liver function based on AST.
Safety of LipoMicel Berberine - Bilirubin | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in liver function based on bilirubin.
Safety of LipoMicel Berberine - Serum creatinine | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in kidney function based on serum creatinine.
Safety of LipoMicel Berberine - Glomerular filtration rate (GFR) | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in kidney function based on GFR.
Safety of LipoMicel Berberine - Fasting blood glucose | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in blood glucose levels based on fasting blood glucose.
Safety of LipoMicel Berberine - Total cholesterol (TC) | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in lipid profile based on TC.
Safety of LipoMicel Berberine - Low-density lipoprotein (LDL) cholesterol | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in lipid profile based on LDL.
Safety of LipoMicel Berberine - High-density lipoprotein (HDL) cholesterol | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in lipid profile based on HDL.
Safety of LipoMicel Berberine - Triglycerides (TG) | 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)
  To evaluate changes in lipid profile based on TG.

SECONDARY OUTCOMES:
Tolerability of Treatment: Bloating | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: Constipation | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: Diarrhea | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: Heartburn | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: cramps | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: knotted feeling in abdomen | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: Rash | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: Nausea | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: Dizziness | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: Blurred vision | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.
Tolerability of Treatment: Other (unrelated to treatment) | From enrollment to the end of treatment at 30 days
  To evaluate tolerability via the collection of health questionnaires. Participants report severity criteria of None, Mild, Moderate, Severe, or Life-threatening.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Solnier, PhD, Principal Investigator — Isura
Locations (1):
- Isura, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No